CLINICAL TRIAL: NCT00944203
Title: Efficacy of Ipomea Pes-caprae Ointment as an add-on Therapy in Patient With Jellyfish Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Watcharapong Piyaphanee, Doctor, Mahidol University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TMEC09-031
Record Dates: First submitted 2009-07-22; First posted 2009-07-23 (Estimated); Last update posted 2018-03-21 (Actual); Status verified 2018-03

CONDITIONS: Jellyfish Dermatitis; Jellyfish Venoms
Keywords: jellyfish; jellyfish venom; jellyfish dermatitis; jellyfish stings; Ipomea pes-caprae

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test Area (Experimental): Test Area = Standard Treatment plus Ipomea pes-caprae oinment
  Interventions: Drug: Ipomea pes-caprae ointment
- Control Area (No Intervention): Control = Standard Treatment

INTERVENTIONS:
Drug: Ipomea pes-caprae ointment — Ipomea pes-caprae ointment will be applied twice a day as an add-on therapy.
  Arms: Test Area

SUMMARY:
This is an open label, prospective, test of superiority efficacy trial of Ipomea pes-caprae ointment as an add-on therapy in patient with jellyfish dermatitis. Each patient will receive standard medical treatment depend on the severity of the disease. The doctor will divide the dermatitis area of each patient into two parts. Ipomea pes-caprae ointment will be applied as an add-on therapy to the "test area", while the ointment will not be applied to the "control area". Patients will be asked to come for follow up 6 times in the 28-days study period. Primary objective is to compare the healing time of dermatitis in both areas.

DETAILED DESCRIPTION:
The "Test area" and "Control area" are allocated in each participant. We use the Internal Control fashion. The healing time of each area will be collected as an outcome measure.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of jellyfish dermatitis
* total lesion area is more than 4 square centimeter

Exclusion Criteria:

* expose to jellyfish more than 7 days
* severe systemic reaction to jellyfish
* allergy to Ipomea pes-caprae or the component of the ointments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2009-07; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Healing time of the Jellyfish dermatitis lesion (days) | Follow up to 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Watcharapong Piyaphanee, MD, Principal Investigator — Mahidol University
Locations (1):
- Hospital for Tropical Diseases, Faculty of Tropical Medicine, Mahidol University, Bangkok, Thailand